CLINICAL TRIAL: NCT04224129
Title: Defining and Quantifying Negative Dysphotopsia Characterization and Causative Factors of Negative Dysphotopsia
Brief Title: Characterization and Causative Factors of Negative Dysphotopsia
Acronym: NDys
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: NDys
Record Dates: First submitted 2017-04-11; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pseudoaphakia
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed as an exploratory study, seeking to investigate the correlation of patient complaints to subjective or objective measurement methods. Better understanding of causative factors of negative dysphotopsia will improve detection and maybe prediction of this optical phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic
* Recurrently and persistently reporting about negative dysphotopsia
* Age 21 and older
* written informed consent prior to entering the study

Exclusion Criteria:

* Relevant ophthalmic diseases such as: glaucoma, (previous) traumatic cataract, corneal scars, age-related macular degeneration and other pathologies resulting in visual field defects
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients after cataract extraction, suffering from negative dysphotopsia
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Identification of factors or a combination thereof that may cause negative dysphotopsia | 2 hours
  Biometry, Anamnesis, visual field, psychological questionnaires, wavefront aberrometry will be used to analyse if a factor causative for negative dysphotopsia can be detected

SECONDARY OUTCOMES:
Method to standardize characterization of negative dysphotopsia | 20 minutes
  New approaches like Goldmann visual field are used to try to picture negative dysphotopsias and patients will also be asked to draw the "dark shadows"
Correlation between eye biometry, patient complaints and psychophysics | 30 minutes
  Eye biometry will be measured using IOL Master 700, patient complaints will be asked during an patient-doctor interview, and psychophysics will be assessed using a psychological questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Prof., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Hanusch-Krankenhaus, Vienna, Austria